CLINICAL TRIAL: NCT03805958
Title: A Randomized Comparison of the Ultrasound-guided Combined Spinal-epidural Anesthesia Technique: Pre-procedure Scan Versus Real-time Scan
Brief Title: Ultrasound-guided Combined Spinal-epidural Anesthesia: Pre-procedure Versus Real-time Scan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 30-2018-81
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Regional Anesthesia Morbidity; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-procedure (Experimental): Confirmed landmark by ultrasound scan before procedure
  Interventions: Procedure: prescan ultrasonography
- Real time (Active Comparator): Confirmed landmark by ultrasound scan during procedure
  Interventions: Procedure: realtime ultrasonography

INTERVENTIONS:
Procedure: realtime ultrasonography — Applying realtime ultrasound during the combined anesthesia
  Arms: Real time
Procedure: prescan ultrasonography — Applying realtime ultrasound before the combined anesthesia
  Arms: Pre-procedure

SUMMARY:
The investigators will compare the success rate, the consumed time, the number of needle passing, the depth and angle of the needle, the anesthetic effect, complications, pain and patient's satisfaction between 'Real-time scan' and 'Pre-procedure scan', when we performing spinal/epidural combined anesthesia.

DETAILED DESCRIPTION:
Traditionally, spinal/epidural combined anesthesia has been performed by palpation of the landmark like Tuffier's line. There are some studies that using ultrasound improves the success rate to regional anesthesia. There are two methods of using ultrasonography, 'Real-time scan' and 'Pre-procedure scan'. Direct comparison of these two methods is not yet studied. So investigators will compare the success rate, the consumed time, the number of needle passing, the depth and angle of the needle, the anesthetic effect, complications, pain and patient's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Spinal/Epidural combined anesthesia is required.

Exclusion Criteria:

* Skin infection or trauma
* Abnormal coagulation lab
* History of spine surgery
* Pregnancy
* Abnormal structure of spine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of needle pass | intraoperative
  Number of needle pass

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyong Kim, Kim, Study Director — SMG-SNU Boramae hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grau T, Leipold RW, Conradi R, Martin E, Motsch J. Ultrasound imaging facilitates localization of the epidural space during combined spinal and epidural anesthesia. Reg Anesth Pain Med. 2001 Jan-Feb;26(1):64-7. doi: 10.1053/rapm.2001.19633. No abstract available. PMID 11172514
- [Background] Kil HK, Cho JE, Kim WO, Koo BN, Han SW, Kim JY. Prepuncture ultrasound-measured distance: an accurate reflection of epidural depth in infants and small children. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):102-6. doi: 10.1016/j.rapm.2006.10.005. PMID 17350519